CLINICAL TRIAL: NCT01479452
Title: Effects of Bariatric Surgery in Swedish Obese Subjects
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOS-1987
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
Keywords: obesity; bariatric surgery; weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bariatric surgery (Other): Bariatric surgery
  Interventions: Procedure: Bariatric surgery
- Controls (Other): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Procedure: Bariatric surgery — Gastric banding, vertical banded gastroplasty, gastric bypass
  Arms: Bariatric surgery
Other: Usual care — Non-surgical obesity treatment
  Arms: Controls

SUMMARY:
The purpose of the Swedish Obese Subjects (SOS) study is to examine the long-term effects of bariatric surgery on overall mortality and obesity-related co-morbidities.

DETAILED DESCRIPTION:
The Swedish Obese Subjects (SOS) study is a prospective non-randomized controlled intervention study designed to examine the long-term effects of bariatric surgery compared to usual care in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 37-60 years and BMI ≥34 kg/m2 in men and ≥38 kg/m2 in women.

Exclusion Criteria:

* Exclusion criteria of both groups were: earlier operation for gastric or duodenal ulcer; earlier bariatric surgery
* Gastric ulcer during the past 6 months; ongoing malignancy
* Active malignancy during the past 5 years
* Myocardial infarction during the past 6 months
* Bulimic eating pattern; drug or alcohol (>0·75 L 40% liquor per week or corresponding amount of ethanol) abuse
* Psychiatric or cooperative problems contraindicating bariatric surgery
* Other contraindicating conditions (such as continuous glucocorticoid or anti-inflammatory treatment).

Ages: 37 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4047 (Actual)
Dates: Start 1987-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 10 years
  The SOS study was started in 1987 and effect of bariatric surgery on overall mortality (primary endpoint) was reported in 2007. Cut off date for the analysis was November 1, 2005.

CONTACTS AND LOCATIONS:
Overall Officials: Lena MS Carlsson, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- SOS secretariat, Vita Straket 15, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Result] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Result] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Result] Sjostrom L, Gummesson A, Sjostrom CD, Narbro K, Peltonen M, Wedel H, Bengtsson C, Bouchard C, Carlsson B, Dahlgren S, Jacobson P, Karason K, Karlsson J, Larsson B, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on cancer incidence in obese patients in Sweden (Swedish Obese Subjects Study): a prospective, controlled intervention trial. Lancet Oncol. 2009 Jul;10(7):653-62. doi: 10.1016/S1470-2045(09)70159-7. Epub 2009 Jun 24. PMID 19556163
- [Derived] Sjoholm K, Svensson PA, Andersson-Assarsson JC, Jacobson P, Ahlin S, Karlsson C, Carlsson B, Kristensson FM, Karlsson P, Peltonen M, Carlsson LMS, Taube M. Sex-specific associations between surgery-induced weight loss and cancer outcomes: A post hoc analysis of the prospective, controlled Swedish Obese Subjects study. PLoS Med. 2026 Jan 5;23(1):e1004876. doi: 10.1371/journal.pmed.1004876. eCollection 2026 Jan. PMID 41490246
- [Derived] Carlsson LM, Peltonen M, Jacobson P, Andersson-Assarsson JC, Svensson PA, Taube M, Karlsson C, Ahlin S, Kristensson FM, Perkins R, Arnetorp I, Carlsson A, Admeus L, Langegard E, Carlsson B, Sjoholm K. Possible selection bias in register-based obesity studies. Eur J Epidemiol. 2025 Jul;40(7):759-766. doi: 10.1007/s10654-025-01237-6. Epub 2025 May 12. PMID 40353980
- [Derived] Carlsson LMS, Arnetorp I, Andersson-Assarsson JC, Jacobson P, Svensson PA, Taube M, Ahlin S, Kristensson FM, Karason K, Larsson I, Karlsson C, Pietilainen KH, Naslund I, Carlsson B, Peltonen M, Sjoholm K. Health outcomes and their association with weight regain after substantial weight loss in Sweden: a prospective cohort study. Lancet Reg Health Eur. 2025 Mar 13;52:101261. doi: 10.1016/j.lanepe.2025.101261. eCollection 2025 May. PMID 40166366
- [Derived] Carlsson LMS, Carlsson B, Jacobson P, Karlsson C, Andersson-Assarsson JC, Kristensson FM, Ahlin S, Svensson PA, Taube M, Naslund I, Karason K, Peltonen M, Sjoholm K. Mortality in relation to diabetes remission in Swedish Obese Subjects - a prospective cohort study. Int J Surg. 2024 Oct 1;110(10):6581-6590. doi: 10.1097/JS9.0000000000001807. PMID 38896851
- [Derived] Kristensson FM, Andersson-Assarsson JC, Peltonen M, Jacobson P, Ahlin S, Svensson PA, Sjoholm K, Carlsson LMS, Taube M. Breast Cancer Risk After Bariatric Surgery and Influence of Insulin Levels: A Nonrandomized Controlled Trial. JAMA Surg. 2024 Aug 1;159(8):856-863. doi: 10.1001/jamasurg.2024.1169. PMID 38748431
- [Derived] Sjoholm K, Andersson-Assarsson JC, Kristensson FM, Hjorth S, Garelius HG, Jacobson P, Svensson PA, Ahlin S, Carlsson B, Peltonen M, Carlsson LMS, Taube M. Long-term incidence of haematological cancer after bariatric surgery or usual care in the Swedish Obese Subjects study: a prospective cohort study. Lancet Healthy Longev. 2023 Oct;4(10):e544-e551. doi: 10.1016/S2666-7568(23)00141-1. Epub 2023 Sep 13. PMID 37716360
- [Derived] Lohmander LS, Peltonen M, Andersson-Assarsson JC, Maglio C, Sjoholm K, Taube M, Jacobson P, Svensson PA, Carlsson LMS, Ahlin S. Bariatric surgery, osteoarthritis and arthroplasty of the hip and knee in Swedish Obese Subjects - up to 31 years follow-up of a controlled intervention study. Osteoarthritis Cartilage. 2023 May;31(5):636-646. doi: 10.1016/j.joca.2022.11.015. Epub 2023 Feb 6. PMID 36754250
- [Derived] Sjoholm K, Carlsson LMS, Svensson PA, Andersson-Assarsson JC, Kristensson F, Jacobson P, Peltonen M, Taube M. Association of Bariatric Surgery With Cancer Incidence in Patients With Obesity and Diabetes: Long-term Results From the Swedish Obese Subjects Study. Diabetes Care. 2022 Feb 1;45(2):444-450. doi: 10.2337/dc21-1335. PMID 34799430
- [Derived] Johansson K, Svensson PA, Soderling J, Peltonen M, Neovius M, Carlsson LMS, Sjoholm K. Long-term risk of anaemia after bariatric surgery: results from the Swedish Obese Subjects study. Lancet Diabetes Endocrinol. 2021 Aug;9(8):515-524. doi: 10.1016/S2213-8587(21)00141-8. Epub 2021 Jul 1. PMID 34217404
- [Derived] Sjoholm K, Jacobson P, Taube M, Svensson PA, Andersson Assarsson JC, Carlsson LMS, Peltonen M. Long-term incidence of hypoglycaemia-related events after bariatric surgery or usual care in the Swedish Obese Subjects study: A register-based analysis. Diabetes Obes Metab. 2021 Aug;23(8):1917-1925. doi: 10.1111/dom.14420. Epub 2021 May 25. PMID 33961331
- [Derived] Taube M, Peltonen M, Sjoholm K, Palmqvist R, Andersson-Assarsson JC, Jacobson P, Svensson PA, Carlsson LMS. Long-term incidence of colorectal cancer after bariatric surgery or usual care in the Swedish Obese Subjects study. PLoS One. 2021 Mar 25;16(3):e0248550. doi: 10.1371/journal.pone.0248550. eCollection 2021. PMID 33764991
- [Derived] Carlsson LMS, Sjoholm K, Jacobson P, Andersson-Assarsson JC, Svensson PA, Taube M, Carlsson B, Peltonen M. Life Expectancy after Bariatric Surgery in the Swedish Obese Subjects Study. N Engl J Med. 2020 Oct 15;383(16):1535-1543. doi: 10.1056/NEJMoa2002449. PMID 33053284
- [Derived] Jacobson P, Peltonen M, Svensson PA, Taube M, Andersson-Assarsson JC, Sjoholm K, Bouchard C, Carlsson B, Carlsson LMS. 9p21.3 Coronary Artery Disease Locus Identifies Patients With Treatment Benefit From Bariatric Surgery in the Nonrandomized Prospective Controlled Swedish Obese Subjects Study. Circ Genom Precis Med. 2020 Oct;13(5):460-465. doi: 10.1161/CIRCGEN.120.003113. Epub 2020 Sep 15. PMID 32931306
- [Derived] Sjoholm K, Carlsson LMS, Taube M, le Roux CW, Svensson PA, Peltonen M. Comparison of Preoperative Remission Scores and Diabetes Duration Alone as Predictors of Durable Type 2 Diabetes Remission and Risk of Diabetes Complications After Bariatric Surgery: A Post Hoc Analysis of Participants From the Swedish Obese Subjects Study. Diabetes Care. 2020 Nov;43(11):2804-2811. doi: 10.2337/dc20-0157. Epub 2020 Sep 1. PMID 32873586
- [Derived] Zhang Y, Peltonen M, Andersson-Assarsson JC, Svensson PA, Herder C, Rudin A, Carlsson L, Maglio C. Elevated adiponectin predicts the development of rheumatoid arthritis in subjects with obesity. Scand J Rheumatol. 2020 Nov;49(6):452-460. doi: 10.1080/03009742.2020.1753808. Epub 2020 Jul 15. PMID 32667228
- [Derived] Ahlin S, Peltonen M, Sjoholm K, Anveden A, Jacobson P, Andersson-Assarsson JC, Taube M, Larsson I, Lohmander LS, Naslund I, Svensson PA, Carlsson LMS. Fracture risk after three bariatric surgery procedures in Swedish obese subjects: up to 26 years follow-up of a controlled intervention study. J Intern Med. 2020 May;287(5):546-557. doi: 10.1111/joim.13020. Epub 2020 Mar 3. PMID 32128923
- [Derived] Kristensson FM, Andersson-Assarsson JC, Svensson PA, Carlsson B, Peltonen M, Carlsson LMS. Effects of Bariatric Surgery in Early- and Adult-Onset Obesity in the Prospective Controlled Swedish Obese Subjects Study. Diabetes Care. 2020 Apr;43(4):860-866. doi: 10.2337/dc19-1909. Epub 2020 Jan 23. PMID 31974103
- [Derived] Taube M, Peltonen M, Sjoholm K, Anveden A, Andersson-Assarsson JC, Jacobson P, Svensson PA, Bergo MO, Carlsson LMS. Association of Bariatric Surgery With Skin Cancer Incidence in Adults With Obesity: A Nonrandomized Controlled Trial. JAMA Dermatol. 2020 Jan 1;156(1):38-43. doi: 10.1001/jamadermatol.2019.3240. PMID 31664428
- [Derived] Maglio C, Zhang Y, Peltonen M, Andersson-Assarsson J, Svensson PA, Herder C, Rudin A, Carlsson L. Bariatric surgery and the incidence of rheumatoid arthritis - a Swedish Obese Subjects study. Rheumatology (Oxford). 2020 Feb 1;59(2):303-309. doi: 10.1093/rheumatology/kez275. PMID 31321442
- [Derived] Jamaly S, Carlsson L, Peltonen M, Jacobson P, Karason K. Surgical obesity treatment and the risk of heart failure. Eur Heart J. 2019 Jul 1;40(26):2131-2138. doi: 10.1093/eurheartj/ehz295. PMID 31089682
- [Derived] Zentenius E, Andersson-Assarsson JC, Carlsson LMS, Svensson PA, Larsson I. Self-Reported Weight-Loss Methods and Weight Change: Ten-Year Analysis in the Swedish Obese Subjects Study Control Group. Obesity (Silver Spring). 2018 Jul;26(7):1137-1143. doi: 10.1002/oby.22200. Epub 2018 Jun 6. PMID 29873894
- [Derived] Maglio C, Peltonen M, Rudin A, Carlsson LMS. Bariatric Surgery and the Incidence of Psoriasis and Psoriatic Arthritis in the Swedish Obese Subjects Study. Obesity (Silver Spring). 2017 Dec;25(12):2068-2073. doi: 10.1002/oby.21955. PMID 29178583
- [Derived] Manousou S, Carlsson LMS, Eggertsen R, Hulthen L, Jacobson P, Landin-Wilhelmsen K, Trimpou P, Svensson PA, Nystrom HF. Iodine Status After Bariatric Surgery-a Prospective 10-Year Report from the Swedish Obese Subjects (SOS) Study. Obes Surg. 2018 Feb;28(2):349-357. doi: 10.1007/s11695-017-2833-0. PMID 28766267
- [Derived] Kanerva N, Larsson I, Peltonen M, Lindroos AK, Carlsson LM. Changes in total energy intake and macronutrient composition after bariatric surgery predict long-term weight outcome: findings from the Swedish Obese Subjects (SOS) study. Am J Clin Nutr. 2017 Jul;106(1):136-145. doi: 10.3945/ajcn.116.149112. Epub 2017 May 17. PMID 28515062
- [Derived] Anveden A, Taube M, Peltonen M, Jacobson P, Andersson-Assarsson JC, Sjoholm K, Svensson PA, Carlsson LMS. Long-term incidence of female-specific cancer after bariatric surgery or usual care in the Swedish Obese Subjects Study. Gynecol Oncol. 2017 May;145(2):224-229. doi: 10.1016/j.ygyno.2017.02.036. Epub 2017 Mar 1. PMID 28259424
- [Derived] Carlsson LMS, Sjoholm K, Karlsson C, Jacobson P, Andersson-Assarsson JC, Svensson PA, Larsson I, Hjorth S, Neovius M, Taube M, Carlsson B, Peltonen M. Long-term incidence of microvascular disease after bariatric surgery or usual care in patients with obesity, stratified by baseline glycaemic status: a post-hoc analysis of participants from the Swedish Obese Subjects study. Lancet Diabetes Endocrinol. 2017 Apr;5(4):271-279. doi: 10.1016/S2213-8587(17)30061-X. Epub 2017 Feb 23. PMID 28237791
- [Derived] Maglio C, Peltonen M, Neovius M, Jacobson P, Jacobsson L, Rudin A, Carlsson LM. Effects of bariatric surgery on gout incidence in the Swedish Obese Subjects study: a non-randomised, prospective, controlled intervention trial. Ann Rheum Dis. 2017 Apr;76(4):688-693. doi: 10.1136/annrheumdis-2016-209958. Epub 2016 Oct 8. PMID 28076240
- [Derived] Keating C, Neovius M, Sjoholm K, Peltonen M, Narbro K, Eriksson JK, Sjostrom L, Carlsson LM. Health-care costs over 15 years after bariatric surgery for patients with different baseline glucose status: results from the Swedish Obese Subjects study. Lancet Diabetes Endocrinol. 2015 Nov;3(11):855-65. doi: 10.1016/S2213-8587(15)00290-9. Epub 2015 Sep 17. PMID 26386667
- [Derived] Sjoholm K, Pajunen P, Jacobson P, Karason K, Sjostrom CD, Torgerson J, Carlsson LM, Sjostrom L, Peltonen M. Incidence and remission of type 2 diabetes in relation to degree of obesity at baseline and 2 year weight change: the Swedish Obese Subjects (SOS) study. Diabetologia. 2015 Jul;58(7):1448-53. doi: 10.1007/s00125-015-3591-y. Epub 2015 Apr 30. PMID 25924987
- [Derived] Konttinen H, Peltonen M, Sjostrom L, Carlsson L, Karlsson J. Psychological aspects of eating behavior as predictors of 10-y weight changes after surgical and conventional treatment of severe obesity: results from the Swedish Obese Subjects intervention study. Am J Clin Nutr. 2015 Jan;101(1):16-24. doi: 10.3945/ajcn.114.095182. Epub 2014 Nov 12. PMID 25527746
- [Derived] Sjostrom L, Peltonen M, Jacobson P, Ahlin S, Andersson-Assarsson J, Anveden A, Bouchard C, Carlsson B, Karason K, Lonroth H, Naslund I, Sjostrom E, Taube M, Wedel H, Svensson PA, Sjoholm K, Carlsson LM. Association of bariatric surgery with long-term remission of type 2 diabetes and with microvascular and macrovascular complications. JAMA. 2014 Jun 11;311(22):2297-304. doi: 10.1001/jama.2014.5988. PMID 24915261
- [Derived] Neovius M, Narbro K, Keating C, Peltonen M, Sjoholm K, Agren G, Sjostrom L, Carlsson L. Health care use during 20 years following bariatric surgery. JAMA. 2012 Sep 19;308(11):1132-41. doi: 10.1001/2012.jama.11792. PMID 22990272
- [Derived] Carlsson LM, Peltonen M, Ahlin S, Anveden A, Bouchard C, Carlsson B, Jacobson P, Lonroth H, Maglio C, Naslund I, Pirazzi C, Romeo S, Sjoholm K, Sjostrom E, Wedel H, Svensson PA, Sjostrom L. Bariatric surgery and prevention of type 2 diabetes in Swedish obese subjects. N Engl J Med. 2012 Aug 23;367(8):695-704. doi: 10.1056/NEJMoa1112082. PMID 22913680
- [Derived] Romeo S, Maglio C, Burza MA, Pirazzi C, Sjoholm K, Jacobson P, Svensson PA, Peltonen M, Sjostrom L, Carlsson LM. Cardiovascular events after bariatric surgery in obese subjects with type 2 diabetes. Diabetes Care. 2012 Dec;35(12):2613-7. doi: 10.2337/dc12-0193. Epub 2012 Aug 1. PMID 22855732
- [Derived] Burza MA, Pirazzi C, Maglio C, Sjoholm K, Mancina RM, Svensson PA, Jacobson P, Adiels M, Baroni MG, Boren J, Ginanni Corradini S, Montalcini T, Sjostrom L, Carlsson LM, Romeo S. PNPLA3 I148M (rs738409) genetic variant is associated with hepatocellular carcinoma in obese individuals. Dig Liver Dis. 2012 Dec;44(12):1037-41. doi: 10.1016/j.dld.2012.05.006. Epub 2012 Jun 15. PMID 22704398